CLINICAL TRIAL: NCT03863899
Title: Pain Control With Ultrasound-guided Ilioinguinal Iliohypogastric Nerve Block Compared With Local Anesthesia Infiltration in Patients Undergoing Transfemoral Transcatheter Aortic Valve Implantation (TF-TAVI): a Prospective, Randomized Trial
Brief Title: Analgesia in Patients Undergoing Transfemoral Transcatheter Aortic Valve Implantation (TF-TAVI)
Acronym: TF-TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Liudmila Hasak, MD, PhD, Principal Investigator, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 305/2018
Record Dates: First submitted 2018-08-10; First posted 2019-03-05 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Aortic Valve Stenosis
Keywords: Ilioinguinal Iliohypogastric nerve block; local anaesthesia infiltration; ultrasound-guided; pain control
MeSH Terms: conditions — Aortic Valve Stenosis; Agnosia | interventions — Nerve Block; Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve block (Experimental): ultrasound-guided ilioinguinal iliohypogastric nerve block performed by the anaesthesiologist for Transaortic valve implantation (TAVI) insertion with eventual additional intraoperative analgesia (AIA) and/or additional postoperative analgesia (APA)
  Interventions: Procedure: Nerve block; Procedure: TAVI; Drug: Additional intraoperative analgesia; Drug: Additional postoperative analgesia
- Local infiltration (Active Comparator): local anaesthesia infiltration performed by the operator for TAVI insertion with eventual intraoperative additional analgesia (AIA) and/or postoperative analgesia (APA)
  Interventions: Procedure: Local infiltration; Procedure: TAVI; Drug: Additional intraoperative analgesia; Drug: Additional postoperative analgesia

INTERVENTIONS:
Procedure: Nerve block — drug mixture: 10-15 ml 0.5% ropivacaine plus 5 ml 1% lidocaine plus 1 mg dexamethasone plus 50 ug adrenaline
  Other Names: Ultrasound-guided ilioinguinal iliohypogastric nerve block
  Arms: Nerve block
Procedure: Local infiltration — 15-20 ml of mixture of 0.5% bupivacaine and 1% lidocaine (1:1)
  Other Names: Local anesthesia infiltration
  Arms: Local infiltration
Procedure: TAVI — Insertion of an aortic valve prothesis through the aorta accessed through femoral artery
  Other Names: Transaortic valve implantation
Drug: Additional intraoperative analgesia — Administration of any analgesics during the operation
  Other Names: AIA
Drug: Additional postoperative analgesia — Administration of any analgesics within first 24 hours after the operation
  Other Names: APA

SUMMARY:
Ilioinguinal and iliohypogastric (ILIH) nerve blocks are frequently performed for analgesia in inguinal surgery.

The investigators hypothesized that preoperative ultrasound-guided ilioinguinal and iliohypogastric (ILIH) nerve blocks will produce better intraoperative analgesia and less analgesic requirement postoperatively in comparison to commonly used preoperative local infiltration anaesthesia for patients undergoing transfemoral transcatheter aortic valve implantation (TF-TAVI).

DETAILED DESCRIPTION:
It is a prospective, randomized trial.

The patients will be randomized to one of the 2 groups:

Group 1 - NERVE BLOCK. Ultrasound-guided ILIH nerve block will be performed by attending anaesthesiologist.

Group 2 - LOCAL INFILTRATION. Local anaesthetic infiltration of the operative area will be performed by operator.

During surgery patients will receive low-dose propofol infusion in order to achieve conscious sedation level, when indicated.

An extra dose of local anaesthetic drug for infiltration of the surgical field or intravenous fentanyl or/and intravenous paracetamol will be given as rescue analgesics in patients reporting pain sensation.

The patients will be observed for 24 hours. The pain at rest will be assessed using numeric rating scale (NRS 0 -10; 0 = no pain: 10 = max pain imaginable).

On the first postoperative day intravenous analgesics will be given on demand (paracetamol 1 g iv (if NRS <5) and oxycodone 2,5 mg iv (if NRS > or = 5)).

ELIGIBILITY:
Inclusion Criteria:

* patients with aortic valve stenosis referred for TF-TAVI
* using a minimalist approach of local anesthesia or nerve block with conscious sedation

Exclusion Criteria:

* patient's refusal to participate
* allergy to local anaesthetic
* TF-TAVI requiring general anesthesia or surgical cut-down
* patients with major cognitive impairment and inability to assess their pain level in Numerical Rating Scale (NRS).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 24 hours
  The numeric rating scale will be used to determine the intraoperative and postoperative pain intensity levels of the patients. Pain intensity is scored 0-10 (0=no pain, 10=the worst pain imaginable). The pain intensity will be measured at 5 time points intraoperatively (femoral artery cannulation, aortic valve system introduction, aortic valve system removal, vessel closure devices insertion and the end of the operation) and at 2 time intervals postoperatively (0-12 hours and 12-24 hours).

SECONDARY OUTCOMES:
Additional intraoperative analgesia consumption | 24 hours
  Fentanyl and paracetamol consumption during the operation.
Additional postoperative analgesia consumption | 24 hours
  Oxycodone and paracetamol consumption in first 24 hours after the operation
Patient satisfaction with analgesia | 3 days
  Categorical quantification: Yes / No
Intraoperative and postoperative cost calculations | 1 year
  Sum of anesthetics and analgesics administered during operation and within first 24 hours after operation

CONTACTS AND LOCATIONS:
Overall Officials: Romuald Lango, MD, PhD, Study Chair — Department of Cardiac Anaesthesiolgy UCC of Gdansk
Locations (1):
- University Clinical Centre, Gdansk, Poland